CLINICAL TRIAL: NCT03172000
Title: Detection of Helicobacter Pylori in Colonic Tissue in Newly Diagnosed Ulcerative Colitis Patients
Brief Title: Detection of Helicobacter Pylori in Ulcerative Colitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IBD Helicobacter
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Colonoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopy and biopsy (Active Comparator): IBD patients
  Interventions: Diagnostic Test: Colonoscopy and biopsy
- Colonoscopic biopsy (No Intervention): Non IBD patients colonoscopic biopsy

INTERVENTIONS:
Diagnostic Test: Colonoscopy and biopsy — Colonoscopic biopsy were taken from the rectum, the sigmoid, descending, transverse, ascending colon, and the cecum of each patient.
  Arms: Colonoscopy and biopsy

SUMMARY:
Helicobacter pylori (H. pylori) infection is one of the most common infectious diseases in humans.

DETAILED DESCRIPTION:
Several bacterial and viral agents may have a role in the aetiology of IBD. In theory, H. pylori infection could be involved in IBD by inducing alterations in gastric and/or intestinal permeability or by causing immunological derangements resulting in absorption of antigenic material and autoimmunity via various immunological pathways.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ulcerative colitis

Exclusion Criteria:

* Other diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Helicobacter | 6 months
  Number of patients with Helicobacter

CONTACTS AND LOCATIONS:
Overall Officials: Loai Mansour, MD, Principal Investigator — Tanta University Faculty of Medicine; Ferial El-kalla, MD, Principal Investigator — Tanta university Faculty of Medicine; Abdelrahman Kobtan, MD, Study Director — Tanta University Faculty of Medicine; Hanan Soliman, MD, Study Director — Tanta University Faculty of Medicine; Sherief Abd-Elsalam, MD, Study Chair — Tanta University Faculty of Medicine
Locations (1):
- Tanta university - faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided